CLINICAL TRIAL: NCT02980081
Title: Abdominal Plain X-ray in the Emergency Departement: Really Usefull?
Brief Title: Abdominal Plain X-ray in the Emergency Departement
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, Professor, Deputy Chief, University Hospital, Geneva
Other Study IDs: CCER 2016-00104
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Emergencies; Diagnostic Imaging; Abdomen, Acute
MeSH Terms: conditions — Emergencies; Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Plain abdominal x-ray: All patients admitted to 2 EDs and with a prescription of an abdominal plain x-ray.
  Interventions: Other: abdominal plain x-ray

INTERVENTIONS:
Other: abdominal plain x-ray — Abdominal plain x-ray as prescribed by the emergency physician

SUMMARY:
There are only few recognized indications for the realization of plain abdominal X-rays in the emergency departement.

The objective of this study is to explore the reasons for abdominal plain X-rays prescription in the Emergency departments (EDs) of two hospitals.

DETAILED DESCRIPTION:
All abdominal plain x-rays prescription will be reviewed in order to identify reasons for prescribing this exam. The indications will be compared to international guidelines in order to identify whether abdominal plain x-rays are overprescribed. Reasons for overprescription will be identify by chart review.

ELIGIBILITY:
Inclusion Criteria:

* >= 16 years
* prescription of an abdominal plain x-ray during their stay in the ED

Exclusion Criteria:

* < 16 y
* no abdominal plain x-ray prescribed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients during one year in 2 EDs in the state of Geneva, Switzerland, with a prescription of an abdominal plain x-ray
Sampling Method: Non-Probability Sample
Enrollment: 1997 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Indications for abdominal plain x-ray prescription | Within 24 hours after ED admission
  Identification of the indications for abdominal plain x-ray and of the number of patients with appropriate indications accordingly to international guidelines

SECONDARY OUTCOMES:
Number and types of other prescribed radiological exams | Within 24 hours after ED admission
  Describe whether other radiological exams (CT, ultrasonography, MRI) have been performed and their indications.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Kherad, MD, MPH, Principal Investigator — Hopital de La Tour
Locations (1):
- Geneva University Hospitals, ED, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertin CL, Ponthus S, Vivekanantham H, Poletti PA, Kherad O, Rutschmann OT. Overuse of plain abdominal radiography in emergency departments: a retrospective cohort study. BMC Health Serv Res. 2019 Jan 14;19(1):36. doi: 10.1186/s12913-019-3870-2. PMID 30642302